CLINICAL TRIAL: NCT06555536
Title: Prospective Study Using the Telemedicine and e-Health Care Method for Patients With Osteogenesis Imperfecta
Brief Title: e-Health Care Method for Patients With Osteogenesis Imperfecta (Tele OI)
Acronym: Tele OI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulo Humberto Mem Martendal Vallandro Costa (Other)
Responsible Party: Sponsor-Investigator, Paulo Humberto Mem Martendal Vallandro Costa, Principal Investigator, Santa Casa de São Paulo
Organization: Santa Casa de São Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCSP
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Intervention Model Description: This is an Interventional Clinical Trial without a Control Group that was carried out in a population of patients with Osteogenesis Imperfecta.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine and e-Health care method for patients with Osteogenesis Imperfecta. (Experimental): This study seeks to formalize the association between the use of technology and the effective treatment of patients with Osteogenesis Imperfecta, not yet explored in the literature.
  Interventions: Other: Tele OI

INTERVENTIONS:
Other: Tele OI — A data collection and Telemedicine tool translated into an APP.

SUMMARY:
This work seeks to formalize the association between the use of technology and the effective treatment of patients with Osteogenesis Imperfecta, which has not yet been explored in the literature; and aims to prove functional improvement in patients, using the MIF scale (Functional Independence Measure) and telemedicine care in addition to telephysiotherapy; to reduce the cost of treatment, allowing the patient to be treated without leaving their home and bringing greater effectiveness to the follow-up of these patients.

DETAILED DESCRIPTION:
This is an Interventional Clinical Trial without a Control Group that was carried out in a population of patients with Osteogenesis Imperfecta. To implement this intervention in these patients, a period of 18 months was required to develop the two pillars that support it: a data collection tool and Telemedicine translated into a dedicated APP, and a YouTube channel with visual guidelines for strengthening exercises and immobilization for possible fractures. The tool was developed through the use of computer programming language (more specifically JavaScript) and today translates into a data collection platform, in addition to also being the virtual environment where participants receive physiotherapy guidance and where they report emergency situations receiving pre-hospital care.

The first consultation of all participants, in accordance with resolution 2227/2018 of the Federal Council of Medicine in Brazil, was carried out in person and all telemedicine care was provided within the outpatient clinics of the Orthopedics Department of Santa Casa de São Paulo, since the records in the medical records were made in the institution's electronic medical record (Soul MV). The intervention began on October 20, 2022 and data were collected until October 20, 2023, although the project remained active and collecting new data due to its success in terms of outcomes. During this period, multidisciplinary monitoring was carried out, being monthly with the orthopedic doctor and the physiotherapist in a digital and synchronous manner. This monitoring was changed only in the case of fractures.

During the follow-up over the almost one-year period of the intervention, the investigators prescribed digital physiotherapy, suggesting that participants perform the activities at least 3 times a week asynchronously (a demand met by almost all). The investigators carry out multidisciplinary consultations via telemedicine every 3 months, changing physiotherapy training within this period to change the stimulation given to the muscles.

ELIGIBILITY:
Inclusion Criteria:

* Osteogenesis Imperfecta patients
* Patients over 3 years old
* Patients must have a smartphone with the possibility of internet access and the capacity to support the Google Meet program (used in teleconsultations).

Exclusion Criteria:

* Patients under 3 years of age
* Patients without any access to any type of internet
* Patients undergoing treatment with pamindronate
* Patients who, due to their older age (above 60 years), were not familiar with a cell phone device to use our application and follow the therapy remotely

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Change Functional Independence Measure (FIM) in OI patients using e-Health | 1 year
  Demonstrate functional improvement of patients, using the FIM scale (Functional Independence Measure) before and after 1 year of intervention using telemedicine care in addition to telephysiotherapy remotely. This scale (FIM) ranges from 7 (minimum and worse outcome) to 126 (maximum and better outcome) and includes measures of independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition. The tool (FIM) is used to assess a patient's level of disability as well as a change in patient status in response to rehabilitation or medical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa de São Paulo, São Paulo, São Paulo, Brazil